CLINICAL TRIAL: NCT07364513
Title: A Phase 1b Open-Label Study of IMSB301 in Subjects With a Type 1 Interferonopathy
Brief Title: Phase 1b Safety Study of IMSB301 in Type 1 Interferonopathies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneSensor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMSB301-101
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Interferonopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMSB301 Treatment (Experimental): IMSB301 Monotherapy
  Interventions: Drug: IMSB301

INTERVENTIONS:
Drug: IMSB301 — Twice daily administration for 28 days.
  Subjects will be treated as out-patient and will return to the clinic at least once weekly on Days 8, 15, 22 and 29.
  Continued treatment beyond Day 28 may be considered on a case-by-case basis for subjects benefiting from treatment.

SUMMARY:
Open-Label Study (Phase Ib) of Type 1 Interferonopathy patients receiving IMSB301 monotherapy.

DETAILED DESCRIPTION:
This is an open-label, Phase Ib study designed to evaluate the safety of IMSB301 monotherapy in Type 1 Interferonopathy patients. The dose of IMSB301 will be based on the recommended Phase Ib dose from Phase Ia.

The following methodology applies to all patients (unless otherwise indicated):

* On Day 1 the first dose of IMSB301 will be administered.
* Subjects will be observed for a minimum period of 6 hours after the dose, and unless acute safety or tolerability issues emerge, they will be discharged and dispensed with study drug sufficient to last until the next visit (Day 8).
* The morning and evening doses will be separated by ~12 hours, and administered at approximately the same time daily.
* Subjects will be treated as out-patients and will return to the clinic at least once weekly. Subsequent study site visits will be morning of Days 8, 15, 22 and 29.
* The subject will have three further visits during the 28-day follow-up period, on Days 36, 43 and 57 (EOS).
* Continued treatment with IMSB301 beyond Day 28 may be considered on a case-by-case basis for subjects benefiting from treatment in the opinion of the Investigator, as outlined in Appendix B.

ELIGIBILITY:
Inclusion Criteria:

1. First subject must be at least 16 years of age and weighing at least 50 kg. Remaining subjects must be at least 12 years of age and weighing at least 40 kg.
2. Molecular diagnosis of one of the following:

   1. Aicardi-Goutières Syndrome (AGS) with mutations in TREX1, RNASEH2A, RNASEH2B, RNASEH2C, SAMHD1, LMS11, or RNU7-11, or
   2. Monogenic SLE with mutations in TREX1, RNASEH2A, RNASEH2B, or RNASEH2C, or
   3. Familial chilblain lupus (CHBL) with mutations in TREX1 or SAMHD1, or
   4. Neurological syndromes with mutations in ATAD3A, or
   5. An unnamed interferonopathy with mutations in DNASE2, or
   6. Coatomer Protein Complex subunit alpha (COPA) syndrome with mutations in COPA. The remaining subtypes of AGS and other type 1 interferonopathies are not eligible.
3. Clinical syndrome consistent with type 1 interferonopathy diagnosis based on clinical, CSF, or radiological findings.
4. Women of child-bearing potential (defined as a female who has experienced menarche and who has not undergone successful surgical sterilization [hysterectomy, bilateral salpingectomy, or bilateral oophorectomy]) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months with an appropriate clinical profile at the appropriate age, e.g., greater than 45 years) must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1.
5. Sexually active male and female subjects with reproductive potential must agree to use highly effective contraception or agree to abstain from heterosexual intercourse throughout the study and for at least 3 months after last study drug dose.
6. Subjects and caregiver must be willing and able to comply with scheduled visits, clinical assessments, blood sample collections, and other trial procedures.
7. Have the ability to provide informed consent or have legal representative of minor/vulnerable subjects who is willing and able to provide written informed consent, provided that assent is obtained from subjects at an age-appropriate level.

Exclusion Criteria:

1. Presence of other significant neurological disorder that is not related to type 1 interferonopathy, brain tumor or other space-occupying lesion, or history of severe head injury.
2. The presence of significant concomitant disease that would, in the judgement of the Investigator, pose additional risk to the subject, interfere with the assessment of safety and tolerability, or significantly interfere with the metabolic disposition of study drug.
3. BMI above 33 kg/m2 or a total body weight in excess of 130 kg.
4. Have any of the following infection risks:

   1. Evidence of active infection during screening or on Day 1
   2. Symptomatic herpes zoster infection within 12 weeks prior to the screening period, or more than one episode of herpes zoster infection in the preceding two years
   3. Positive hepatitis B, hepatitis C, HIV or TB test at screening
   4. Household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB
   5. Serious infection, defined as infection requiring admission to hospital or treatment with intravenously administered medication, within the six months.
5. Resting 12-lead ECG showing confirmed prolongation of QTc (Fridericia's correction) interval (QTc interval > 470 for females and >450 for males), or other baseline ECG abnormalities that, in the judgement of the Investigator, would pose additional safety risk to the subject.
6. A prior history of cancer, other than squamous cell carcinoma, basal cell carcinoma, or cervical intra-epithelial neoplasia that was successfully treated at least five years prior to the screening visit and which has shown no sign of clinical recurrence.
7. Receipt of an investigational drug within 30 days or five half-lives of the drug (whichever is longer) prior to Day -1.
8. Prior treatment with an immunomodulator including a JAK inhibitor within 14 days of screening.
9. Prior treatment with an interferon inhibitor within 3 months of screening.
10. Concurrent treatment of a nucleoside reverse transcriptase inhibitor or other antiviral drug.
11. Receipt of a strong inhibitor of CYP3A4 (APPENDIX A) within five half-lives prior to Day -1
12. Known allergy to IMSB301 or its components.
13. Known allergy to shellfish.
14. Female subjects who are breastfeeding or who have a positive pregnancy test at screening or Day -1.
15. Receipt of a vaccination within 3 weeks prior to Day -1.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Drug-related safety | 57 days
  Incidence of subjects with Adverse Events

SECONDARY OUTCOMES:
Target engagement as measured by Pharmacokinetics | 29 Days
  Peak plasma concentration (Cmax)
Target engagement as measured by Pharmacokinetics | 29 Days
  Trough plasma concentration (Cmin)
Target engagement as measured by Pharmacokinetics | 29 Days
  Area under the plasma concentration versus time curve (AUC)
Target engagement as measured by Pharmacodynamics | 43 Days
  Changes to interferon score based on 6 interferon signature gene (ISG) expression levels in whole blood
Target engagement as measured by Pharmacodynamics | 43 Days
  Determination of interferon alpha (IFNa) protein levels in plasma
Target engagement as measured by Pharmacodynamics | 43 Days
  Changes to Interferon beta (IFNb) expression levels in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital at Westmead, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No